CLINICAL TRIAL: NCT06635252
Title: Statins, Cholesterol and Cognitive Decline in Alzheimer's
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Sara Garcia-Ptacek, Assistant Professor | Docent, Karolinska Institutet
Other Study IDs: 2024-00178-02
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer Dementia; Statins
MeSH Terms: conditions — Alzheimer Disease | interventions — elesclomol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Alzheimer's disease: Prospective cohort study based on data from the Stockholm Creatinine Measurements (SCREAM) project. Patients diagnosed with AD and mixed dementia and registered in the Swedish Registry for Cognitive/Dementia Diseases are included.
  Interventions: Drug: STA 4783

INTERVENTIONS:
Drug: STA 4783 — Use of statins will be identified from Prescribed Drug register within 6 months before dementia diagnosis or each follow-up date

SUMMARY:
Disturbances in brain cholesterol homeostasis may be involved in the pathogenesis of Alzheimer's disease (AD). Lipid-lowering medications could interfere with neurodegenerative processes in AD through cholesterol metabolism or other mechanisms. The investigators aim to estimate the causal effect of statins on cognitive function measured by MMSE and to identify the mediating or modifying effect of cholesterol between statins and cognitive function in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

All patients with AD and mixed dementia registered in SveDem and from SCREAM.

Exclusion Criteria:

* All patients with a missing MMSE score at diagnosis date will be excluded from the analyses.
* Patients with at least one measurement of low-density lipoprotein cholesterol (LDL-C) within 1 year before dementia diagnosis.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort study based on data from the Stockholm Creatinine Measurements (SCREAM) project, linking laboratory data with SveDem-the Swedish Registry for Dementia Cognitive disorders, the National Patient Registry, the Swedish Prescribed Drug Registry, The Swedish Cause of Death Register and Health Insurance and Labour Market Studies (LISA). Dates between May 1, 2007, and October 16, 2018
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Cognitive decline | Through study completion, at least 1 year
  The data on cognitive change will be assessed by Mini Mental State Examination (MMSE) score. The MMSE score ranges from 0 and 30. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No